CLINICAL TRIAL: NCT06725485
Title: Low-Dose Lidocaine Infusion for Acute Pain Management in the Surgical Intensive Care Unit - A Pilot Study
Brief Title: Low-Dose Lidocaine Infusion for Acute Pain Management Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Hina Faisal, Assistant Professor of Clinical Surgery, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00027972
Record Dates: First submitted 2024-11-19; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Pain Management
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Low-Dose Lidocaine Infusion (Experimental): Low-dose lidocaine infusion 10-30 mcg/kg/min administered within 1 hour of ICU admission.
  Interventions: Drug: Low-Dose Lidocaine

INTERVENTIONS:
Drug: Low-Dose Lidocaine — Low-dose lidocaine infusion 10-30 mcg/kg/min administered within 1 hour of ICU admission.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of lidocaine infusion in acute pain management following open abdominal surgery, including opiate use after surgery and the incidence of postoperative nausea and vomiting, Ileus, length of stays (ICU/hospital), and improvement in patient satisfaction.

DETAILED DESCRIPTION:
The management of acute pain remains challenging for the physicians, with many patients suffering from inadequate pain control following surgery. Evidence has shown that 90% of patients in the intensive care unit usually treated with opioids for pain. Poorly controlled pain and opioid-related adverse events have several negative consequences for critically ill patients during the postoperative period, including delay in functional recovery and hospital discharge, increased length of stay, development of chronic postsurgical pain, reduced patient satisfaction, and increased total healthcare cost. The reported incidence of postoperative Ileus varies with the procedure, ranging from 14.9% for large-bowel resection and 19.2% for small-bowel resection). Although many analgesic therapies are available, the high incidence of postoperative pain among patients indicates that there are still significant treatment challenges. Recently, there has been much interest in using low-dose lidocaine infusion for acute pain management in the operating room or/and PACU. Lidocaine is a drug with multiple effects, including anti-arrhythmic, local, topical, and injectable anesthetics. Lidocaine is also used for uncontrolled and chronic pain. However, this is an off-label use. Additionally, I.V. lidocaine is a potent anti-inflammatory, anti-hyperalgesic, and gastrointestinal pro-peristaltic drug. There is a lack of data on low dose lidocaine infusion for acute postoperative pain management in surgical critical care patients.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age > 18 years admitted to surgical ICU.
* Severe acute pain with pain scale > 7, following open exploratory laparotomy for bowel, gall bladder, and pancreatic surgeries.
* Women of childbearing age must have a negative urine/serum pregnancy test.

Exclusion Criteria:

* Regional anesthesia during surgery
* Heart failure with ejection fraction < 20%.
* Allergy to amide local anesthetics
* Neuraxial anesthesia during surgery
* Post-liver transplant patients
* Hemodynamically unstable patients on two or more vasopressors
* Child-Pugh Class C or MELD >20
* Any investigational drug use within 30 days before enrollment
* Pregnant or lactating females
* Patients with chronic opioid-dependence
* Intubated and mechanically ventilated patients on intensive care unit analgo-sedation
* Subjects who do not agree to participate or may be non-compliant with study schedules or procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Opioid consumption on post-operative day 3 | Post-operative day 3
  Opioid consumption in a 24-hour period starting 3 days after surgery, measured in morphine milligram equivalents

SECONDARY OUTCOMES:
Pain Scale at 72 Hours Post-Surgery | Post-operative day 3
  Patient numeric pain scale rating (0-10), with 0 being no pain and 10 being the worst pain possible
Opioid-Free Days | Time of surgery through the end of post-operative day 3
  The proportion of days post-surgery that the patient did not require opioid analgesia
Time Until Return in bowel function | Time of surgery through discharge, up to 30 days
  Post-operative day when patient first has a bowel movement
Return to Oral Feeding | Time of surgery through discharge, up to 30 days
  Post-operative day number when patient returns to oral feeding
Post-operative intensive care unit length of stay | Time of surgery through intensive care unit discharge, up to 1 year
  Number of days between surgery and discharge from the intensive care unit after surgery
Post-operative hospital length of stay | Time of surgery through hospital discharge, up to 1 year
  Number of days between surgery and discharge from hospital after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No